CLINICAL TRIAL: NCT05910229
Title: Interest of a Telephone Paramedical Support Prior to the Radiotherapy Simulation Scanner to Ensure the Realization of Specific Recommendations for the Management of Patients with Prostate Cancer.
Brief Title: Telephone Paramedical Support Prior to the Radiotherapy Simulation Scanner for Patients with Prostate Cancer
Acronym: RTEPROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de Bretagne Sud (Other)
Responsible Party: Principal Investigator, Rosalie Guegan, Principal Investigator, Groupe Hospitalier de Bretagne Sud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 56LORC_2021_RTEPROST
Record Dates: First submitted 2023-05-05; First posted 2023-06-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Radiotherapy; Prostate Cancer
Keywords: paramedical phone call
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: comparative monocentric study with randomisation between two parallel arms
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient with standard care (No Intervention): Consultation with the onco radiotherapeutic and submission of the recommendations to follow before the simulation CT Scan before the radiotherapy
- Patient with personalized support (Experimental): Consultation with the onco radiotherapeutic and submission of the recommendations to follow before the simulation CT Scan before the radiotherapy and a phone call by a radiotherapy technician
  Interventions: Other: Phone call

INTERVENTIONS:
Other: Phone call — In the experimental arm the patient will be called 3 days before the CT scan
  Arms: Patient with personalized support

SUMMARY:
The goal of this clinical trial is to evaluate the impact of a phone call before the simulation CT scan in management of care of patients with prostate cancer.

DETAILED DESCRIPTION:
After being informed about the study, all patients who have given written informed consent and who met eligibility requirement will be randomized in a simple blind manner ( investigator) in a 1:1 ration.

The main question it aims to answer is : Does a phone call before the simulation CT scan has an effectiveness on patients compliance of the recommendations and therefore on obtaining quality images.

There is no additional risk of patients involvement.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Patient coming for prostate cancer treatment with or without lymph node irradiation
* Minimum of 48 hours between the onco radiotherapist and the CT scan
* Signed a written informed consent form
* Affiliated to the social security system

Exclusion Criteria:

* Patient not understanding French
* Patient not reachable by phone
* Individual of full age deprived of liberty or placed under a legal protection measure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Assess the value of a telephone call in terms of compliance recommendations for preparation (empty rectum and full bladder) necessary to perform the CT scanner simulation in the management of patients with prostate cancer. | From the day of the consultation with the radiotherapist to the day of the CT scanner, up to three month after the inclusion
  The proportion of patients for whom it is necessary to renew the CT scanner simulation.

SECONDARY OUTCOMES:
Assess the impact of a telephone call upstream of the simulation scanner on patient preparation according to recommendations. | From the day of the consultation with the radiotherapist to the day of the CT scanner, up to three month after the inclusion
  The number of patients who performed the preparation for the scanner.
Assess the impact of a telephone call upstream of the simulation scanner on reading the recommendation sheet given to the patient during the announcement medical consultation. | From the day of the consultation with the radiotherapist to the day of the CT scanner, up to three month after the inclusion
  The number of patients who read the recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Rosalie GUEGAN, Principal Investigator — GHBretagne sud
Locations (1):
- Hôpital du Scorff, Lorient, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Crevoisier R, Tucker SL, Dong L, Mohan R, Cheung R, Cox JD, Kuban DA. Increased risk of biochemical and local failure in patients with distended rectum on the planning CT for prostate cancer radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):965-73. doi: 10.1016/j.ijrobp.2004.11.032. PMID 15989996
- [Background] Maggio A, Gabriele D, Garibaldi E, Bresciani S, Delmastro E, Di Dia A, Miranti A, Poli M, Varetto T, Stasi M, Gabriele P. Impact of a rectal and bladder preparation protocol on prostate cancer outcome in patients treated with external beam radiotherapy. Strahlenther Onkol. 2017 Sep;193(9):722-732. doi: 10.1007/s00066-017-1163-4. Epub 2017 Jun 15. PMID 28620751